CLINICAL TRIAL: NCT00585286
Title: Evaluation of a Novel Fractional Resurfacing Device for the Treatment of Acne Scarring
Brief Title: Fractional Resurfacing Device for Treatment of Acne Scarring
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Reliant Technologies, Inc. Mountain View, CA (Industry); University of Minnesota (Other)
Responsible Party: Principal Investigator, Christopher Zachary, Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-5328
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Acne; Scar
Keywords: acne vulgaris; scarring; laser
MeSH Terms: conditions — Acne Vulgaris; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fractional carbon dioxide laser system (Experimental): Thirty total healthy subjects from two research centers with skin type I-IV of moderate to severe acne scarring received treatment with the 10,600 nm fractional carbon dioxide laser system.
  Interventions: Device: 10,600 nm fractional carbon dioxide laser system

INTERVENTIONS:
Device: 10,600 nm fractional carbon dioxide laser system — 1-3 laser treatments using 20-100 millijoules (mJ) with 100-400 microscopic treatment zones (MTZ)/cm2 per pass and total density of 600-1200 MTZ/cm2
  Other Names: Fraxel Re:pair laser

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of a new investigational laser device for treatment of acne scarring, for improvement in the appearance of surface texture and topography (recessed or uneven surfaces).

DETAILED DESCRIPTION:
Thirty subjects between two research locations with an acne scar severity score greater than 4 will receive up to 3 treatments with an FDA IDE and Institutional Review Board approved 10,600nm fractional carbon dioxide laser system. Improvement of acne scarring is evaluated at 1 month and 3 months post-treatment.

Post-treatment responses evaluated are immediate erythema, immediate edema, and any other immediate responses. Evaluations are conducted immediate post treatment and one week post-treatment. Key safety data include the severity scoring of post-treatment responses, as well as by photodocumentation.

The incidence of side effects such as scarring, pigmentary changes, etc. are evaluated at follow-up visits one and three months post-treatment. Key safety data include the incidence rates and severity scoring of side effects, as well as by photodocumentation

ELIGIBILITY:
Inclusion Criteria:

* Have Fitzpatrick skin type I-V. (Type I is blonde/red hair with freckles and Type V are Hispanics and lighter African Americans.)
* Are male or female.
* Are between 18 and 75 years of age.
* Have moderate to severe acne scarring. Acne scarring will be assessed with the Acne Scar Severity Scale. Subjects will be eligible for treatment if the area to be treated is scored as having an Acne Scar Severity Score > 4 according to the Acne Scar Severity Scale (0-9).
* Are able to read, understand, and sign the Informed Consent.
* Are willing and able to comply with all follow-up requirements for a minimum of 8 months.

Exclusion Criteria:

* Have had active localized or systemic infections within 6 months of enrollment
* Have compromised ability for wound healing, such as: malnutrition, oral steroid use, history of collagen vascular disease (e.g. lupus, scleroderma, history of keloid formation (raised and thickened scars), atrophic dermatitis (extreme skin irritation or itchiness) or immunologic abnormalities such as vitiligo (white patches of skin due to loss of pigment)
* Have immunocompromised status (inability to resist infection, etc.)
* Have been treated with lasers, chemical procedures, or other cosmetic procedures on the area to be treated within 6 months of enrollment
* Have taken Accutane within 12 months of enrollment
* Are allergic to lidocaine (skin numbing agent)
* Are allergic to Valtrex (an anti-viral medication)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Zachary, MBBS, FRCP, Principal Investigator — University of California, Irvine; Brian D Zelickson, MD, Principal Investigator — Department of Dermatology, University of Minnesota, Minneapolis, Minnesota
Locations (1):
- UC Irvine Dermatology Clinical Research Center, Irvine, California, United States

REFERENCES:
- See also: University of California, Irvine Department of Dermatology Clinical Research — http://www.dermatology.uci.edu/clinical_trials.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 total patients with moderate to severe acne scarring were recruited from 3/2007-5/2008 between two locations. Of these, 15 patients received treatment and 14 patients completed the full course of the study at the University of California, Irvine General Clinical Research Center.
Pre-assignment Details: Subjects must not have been treated with other lasers, chemical procedures, or other cosmetic procedures on the area to be treated within 12 months of enrollment.
Groups:
- Fractional Carbon Dioxide Laser System: Fifteen healthy subjects of skin type I-IV received treatment with the 10,600 nm fractional carbon dioxide laser system.
Period: Overall Study
Arm/Group | Fractional Carbon Dioxide Laser System
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Of 30 patients enrolled between two research centers, 15 subjects were enrolled at the UC Irvine General Clinical Research Center
Groups:
- Fractional CO2 Laser System: Thirty healthy subjects of skin type I-IV received treatment with the 10,600 nm fractional CO2 laser system.
Arm/Group | Fractional CO2 Laser System
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Improvement of Acne Scarring
Description: Subject assessment of the percent improvement of acne scarring compared to baseline and based on the quartile scale (0: no improvement; 1: 1-25% improvement; 2: 26-50%; 3: 51-75%; 4: 76-100% improvement).
Time Frame: Baseline, 1 month and 3 months post-treatment
Population: Out of 15 subjects enrolled at our site, one was lost to follow up before the 3 month follow up for the first treatment. Therefore, data was analyzed for the 14 patients that completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fractional CO2 Laser System: Fifteen healthy subjects of skin type I-IV received treatment with the 10,600 nm fractional CO2 laser system.
Arm/Group | Fractional CO2 Laser System
Number analyzed (Participants) | 14
units on a scale
  Month 1 | 2.26 (1.15)
  Month 3 | 1.91 (1.0)

2. Primary Outcome: Average Improvement in Surface Texture
Description: Subject assessment of the percent improvement of surface texture compared to baseline and based on the quartile scale (0: no improvement; 1: 1-25% improvement; 2: 26-50%; 3: 51-75%; 4: 76-100% improvement).
Time Frame: Baseline, 1 month and 3 months post-treatment
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Fractional CO2 Laser System
Number analyzed (Participants) | 14
units on a scale
  Month 1 | 1.94 (1.16)
  Month 3 | 2.09 (0.85)

3. Primary Outcome: Degree of Atrophy
Description: Subject assessment of the percent improvement in extent of atrophy compared to baseline and based on the quartile scale (0: no improvement; 1: 1-25% improvement; 2: 26-50%; 3: 51-75%; 4: 76-100% improvement).
Time Frame: Baseline, 1 month and 3 months post-treatment
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Fractional CO2 Laser System
Number analyzed (Participants) | 14
units on a scale
  Month 1 | 1.68 (1.11)
  Month 3 | 1.65 (1.14)

4. Secondary Outcome: Pain Tolerance
Description: The average pain score reported over all three treatments was 5.67, corresponding to "moderate" pain based on a 10-point scale. The pain score is recorded on a 10-point scale, with 0 being "no pain" and 10 being "worst pain imaginable." All subjects reported that any discomfort associated with the procedure was only during active intervention and resolved immediately post-procedure. Increased pain scores correlated with increased density, but not increased energy.
Time Frame: At treatment visit (up to 3 visits)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fractional CO2 Laser System
Number analyzed (Participants) | 14
units on a scale | 5.67 (0.833)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire study for approximately 1 year and 3 months.
Arm/Group | Fractional CO2 Laser System
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
There were no major limitations to this trial. The trial was completed without any technical problems or major complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No